CLINICAL TRIAL: NCT07285161
Title: Evaluating the Impact of a Positive Health Dialogue Tool in Veterans With PTSD: A Randomised Controlled Trial
Acronym: EIPHDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reinier van Arkel (Other)
Responsible Party: Principal Investigator, Maarten Muskens, Drs., Reinier van Arkel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RvA_PTCZN_NL72664.068.20; NL72664.068.20 (Other: METc Maastricht University)
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: Veterans; Post Traumatic Stress Disorder; Positive Health; Recovery; Randomised Controlled Trial
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Forty-four veterans diagnosed with PTSD were randomly assigned to either a treatment group, which received two additional sessions using the dialogue tool alongside standard trauma-focused therapy, or a control group receiving treatment as usual.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Positive Health dialogue tool
  Interventions: Behavioral: Positive Health dialogue tool
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Positive Health dialogue tool — This intervention is distinguished by the integration of a structured dialogue tool in two additional sessions, designed to enhance therapeutic engagement and reflection. Unlike standard trauma-focused therapy alone, this approach offers a unique combination of conventional treatment with a targeted communication strategy tailored to veterans with PTSD.
  Arms: Intervention group

SUMMARY:
The primary outcome is quality of life, with secondary outcomes including PTSD symptoms, and psychosocial functioning. We hypothesise that a low-dose intervention based on empowerment and self-directed goal setting will lead to (a) measurable improvements in veterans' quality of life and (b) reduced PTSD symptoms, and improved psychosocial functioning.

DETAILED DESCRIPTION:
Background: Veterans with post-traumatic stress disorder (PTSD) often experience complex and persistent symptoms that extend beyond the scope of trauma-focused treatments. The Positive Health framework offers an integrative approach to health and well-being, yet its application in veteran populations remains unexplored. This randomized controlled trial investigated the effects of integrating the Positive Health dialogue tool into trauma-focused treatment for veterans with PTSD. The study aimed to evaluate its impact on recovery indicators, including quality of life, PTSD symptoms, and psychosocial functioning. Methods: Forty-four veterans diagnosed with PTSD were randomly assigned to either a treatment group, which received two additional sessions using the dialogue tool alongside standard trauma-focused therapy, or a control group receiving treatment as usual. Outcomes were measured at baseline, 6 months, and 12 months using validated instruments, including the MANSA, PCL-5, and TRACK 2.0. Results: Although both groups showed improvements over time in PTSD symptoms and psychosocial functioning, there were no statistically significant differences found between the treatment and control groups across various recovery indicators. Conclusions: The limited scope, lack of iintegration, and timing of the intervention may have contributed to the absence of measurable effects. While the dialogue tool did not yield additional benefits beyond standard treatment, the findings underscore the need for more structured, integrated, and timely recovery-oriented interventions. Trial registration: The study was approved by the Medical Ethics Committee of Maastricht University (METc azM/UM) and registered under number NL72664.068.20 on July 7, 2020. This study was funded by the Dutch National Care System for Veterans (Landelijk Zorgsysteem voor Veteranen, LZV), which supports research aimed at improving mental health care for military veterans in the Netherlands. Corresponding author: Drs. M.M.P.A. (Maarten) Muskens: Psychotraumacentrum Zuid-Nederland; address: Bethaniestraat 10, 5211JL 's- Hertogenbosch, The Netherlands; phone: 0031 73 658 64 00; email: Maarten. Muskens@reiniervanarkel.nl

ELIGIBILITY:
Inclusion Criteria:

* A formal PTSD diagnosis
* At the start of treatment
* Aged 18 until 64
* Reading, writing, and speaking Dutch

Exclusion Criteria:

* Alcohol or drug dependency
* Severe cognitive impairments (e.g., dementia)
* Acute suicide risk, as assessed during the intake procedure

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life Scores from Baseline, 6 Months, and 12 Months as Measured by the MANSA Questionnaire | From enrollment to 12 months post-enrollment

SECONDARY OUTCOMES:
Change in PTSD Symptom Severity from Baseline, 6 Months, and 12 Months as Measured by the PCL-5 Questionnaire | rom enrollment to 12 months post-enrollment
Change in Psychosocial Functioning from Baseline, 6 Months, and 12 Months as Measured by the TRACK 2.0 Questionnaire | From enrollment to 12 months post-enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier van Arkel, Psychotraumacentrum Zuid-Nederland, 's-Hertogenbosch, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study will be stored in a nonpublicly available repository en will be available upon request from the corresponding author.